CLINICAL TRIAL: NCT01928381
Title: A Randomized, Double-Blind, Placebo-Controlled Crossover Study to Evaluate the Preliminary Efficacy of AZD5213 in Combination With Pregabalin in Subjects With Painful Diabetic Neuropathy and Good Pain Reporting Ability
Brief Title: Safety, Tolerability and Preliminary Efficacy of AZD5213 in Combination With Pregabalin in Subjects With PDN and Good Pain Reporting Ability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3031C00001
Record Dates: First submitted 2013-08-21; First posted 2013-08-23 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Neuropathy, Painful; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo capsules (Placebo Comparator): Capsules to match pregabalin and AZD5213
  Interventions: Drug: Placebo
- AZD5213 + pregabalin (Experimental): AZD5213 in combination with pregabalin
  Interventions: Drug: AZD5213 + pregabalin
- pregabalin (Active Comparator): pregabalin capsules
  Interventions: Drug: pregabalin capsules

INTERVENTIONS:
Drug: AZD5213 + pregabalin — Double blind Investigational drug AZD5213 (capsules) given in combination with pregabalin (capsules)
  Other Names: pregabalin (LYRICA)
  Arms: AZD5213 + pregabalin
Drug: Placebo — Double blind placebo capsules to match AZD5213 and pregabalin
  Arms: placebo capsules
Drug: pregabalin capsules — Double blind pregabalin capsules to match AZD5213 and placebo
  Other Names: LYRICA (pregabalin)
  Arms: pregabalin

SUMMARY:
This is a 2-part study. In Part 1 of the study, subjects will undergo a pain reporting training program in which a painful stimulus will be applied to the subject's hand, and the subjects will be asked to report how painful the stimulus is. Over the course of the pain training sessions, feedback will be provided to the subject about how accurately they are reporting their degree of pain, relative to the amount of pressure stimulus applied to evoke pain. Those subjects who have adequate pain reporting ability will be asked to continue into Part 2 of the study in which 3 different blinded study drugs will be administered to each subject, in a crossover design to compare whether or not the study drugs improve pain associated with diabetic neuropathy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, two-part study in adults (ages 18-75 years) with Painful Diabetic Neuropathy (PDN).

In Part 1 of the study, eligible subjects will enter a 4-week Pain Training Period. During the Pain Training Period, subjects will receive three weekly in-clinic training sessions using repeated rating of experimental pressure pain stimuli. Subjects will receive feedback during this training and will be evaluated on their pain-reporting ability during each in-clinic session. Subjects with acceptable pain-reporting ability at the conclusion of the Pain Training Period will be eligible to enter Part 2 of the study. Subjects with unacceptable pain-reporting ability at the conclusion of the Pain Training Period will be discontinued from the study.

Part 2 of the study will consist of three consecutive double-blind crossover periods. Each crossover period will include 31 days of double-blind treatment. A follow-up visit will occur 14 ± 7 days after the last dose of study medication.

One of three treatments (placebo, pregabalin, or pregabalin + AZD5213) will be administered during each crossover treatment period, as determined by a randomly assigned treatment sequence.

Approximately 65 subjects will be screened in Part 1 of the study, in order to randomize up to approximately 32 subjects in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 75 years, inclusive, at Screen. 2. Subjects must provide informed consent in accordance with local regulations before the conduct of any study-related procedures. The informed consent should reflect the protocol stipulations concerning the use of contraception. 3. Diagnosis of Type 1 or Type 2 diabetes mellitus for at least 1 year prior to Screen. 4. Diabetes-related painful neuropathy for at least 6 months prior to Screen. 5. Pain that began in the feet and is symmetric or nearly symmetric. 6. Diabetes has been clinically stable for at least 2 months prior to Screen, and between Screen and baseline (Day 35). 7. At Screen and baseline, score of at least 4 on Item 5 ("average pain") of the modified Brief Pain Inventory for patients with painful diabetic peripheral neuropathy (BPI-DPN). 8. Able to participate in all scheduled evaluations and to complete all required tests and procedures. 9. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to pregabalin. 2. Clinically important illness or infection (e.g., chronic, persistent, or acute infection) within 30 days prior to screen or between screen adn baseline. 3. Presence of any psychiatric or neurologic disorder or any other disorder or symptom, if, in the judgement of the investigator, the disorder or symptom is likely to confound interpretation of drug effect or affect the subject's ability to complete the study. Any clinically important abnormality, as determined by investigator at Screen or baseline, in physical or neurologic examination, vital sign, ECG, or clinical laboratory test results that could be detrimental to the subject, or could affect the subject's ability to complete the study. 4. Initiation or change in intensity or frequency of non-pharmacologic therapy for PDN, including psychotherapy, physical therapy, massage, acupuncture, acupressure, or chiropractic care, within 3 months prior to baseline).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Clearwater, Florida
  - Research Site, Orlando, Florida
  - Research Site, Newnan, Georgia
  - Research Site, Brockton, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 143 adults with painful diabetic neuropathy were screened, in a total of 146 screenings, 83 met eligibility criteria and entered Pain Training - Part 1. To be randomized into Part 2 (3 period treatment crossover study), participants had to successfully complete Part 1 Pain Training and meet all study entry criteria at Visit 6 (~Day 36) .
Pre-assignment Details: Crossover data starting with First Intervention excludes 3 participants who were randomized but not treated in the double-blind crossover periods. The 3 are included as withdrawals in Part 1 - Placebo run-in (single blind) period.
Groups:
- Part 1 - Pain Training: Part 1 - Screening, Pain Training, placebo run-in eligibility for Part 2
- Sequence 1: Sequence 1 - 1st placebo, 2nd pregabalin, 3rd AZD5213 + pregabalin
- Sequence 2: Sequence 2 - 1st Placebo, 2nd AZD5213 + pregabalin, 3rd pregabalin
- Sequence 3: Sequence 3 - 1st pregabalin, 2nd placebo, 3rd AZD5213 + pregabalin
- Sequence 4: Sequence 4 - 1st pregabalin, 2nd AZD5213 + pregabalin, 3rd placebo
- Sequence 5: Sequence 5 - 1st AZD5213 + pregabalin, 2nd placebo, 3rd pregabalin
- Sequence 6: Sequence 6 - 1st AZD5213 + pregabalin, 2nd pregabalin, 3rd placebo
Period: Screening for Pain Training
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 143 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 83 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 60 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not qualify (inclusion/Exclusion) | 60 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 - Pain Training
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 83 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 48 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pain training criteria not met | 29 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo run-in & Part 2 Eligibility
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 48 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 34 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Eligibility for Part 2 not met | 10 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - First Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 6 | 6 | 6 | 4 | 6 | 6
Completed | 0 | 6 | 4 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 2 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study specific withdrawal criteria | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Eligibility criterion not met | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout First Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 6 | 4 | 5 | 4 | 5 | 5
Completed | 0 | 6 | 4 | 5 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 2 - Second Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 6 | 4 | 5 | 3 | 5 | 5
Completed | 0 | 5 | 4 | 4 | 3 | 5 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 0
Period: Washout Second Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 5 | 4 | 4 | 3 | 5 | 5
Completed | 0 | 5 | 4 | 4 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - Third Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 5 | 4 | 4 | 3 | 5 | 5
Completed | 0 | 5 | 4 | 4 | 3 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - Post Third Intervention
Arm/Group | Part 1 - Pain Training | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 0 | 5 | 4 | 4 | 3 | 5 | 5
Completed | 0 | 5 | 3 | 4 | 3 | 5 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Started Part 1
Groups:
- Overall Study: Overall Study - Starting with Part 1
Arm/Group | Overall Study
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 43
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Index - Item 5, Average Daily Pain Score (Range 0-10) Higher Values Indicate Worse Pain
Description: Brief pain Index - diabetic painful neuropathy (BPI-DPN) - average daily pain, Item 5 (final 2 day diary + in clinic assessment at end of 3 week treatment period)
Time Frame: 3 weeks of treatment
Population: Full Analysis set
Measure: Least Squares Mean (Standard Error); unit: Average daily pain score
Groups:
- Part 2 - Placebo: Part 2 - placebo crossover periods
- Part 2 - Pregabalin + AZD5213: Part 2 - Combined pregabalin + AZD5213 crossover periods
- Part 2 - Pregabalin: Part 2 pregabalin crossover periods
Arm/Group | Part 2 - Placebo | Part 2 - Pregabalin + AZD5213 | Part 2 - Pregabalin
Number analyzed (Participants) | 29 | 27 | 30
Average daily pain score | 4.24 (0.38) | 4.41 (0.38) | 4.27 (0.38)
Statistical Analysis 1: Comparison: Part 2 - Pregabalin + AZD5213 vs Part 2 - Pregabalin; Test type: Superiority or Other; p = 0.5695, Mixed Models Analysis; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.34 to 0.61], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Part 2 - Placebo vs Part 2 - Pregabalin; Test type: Superiority or Other; p = 0.8905, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.43 to 0.49], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Part 2 - Placebo vs Part 2 - Pregabalin + AZD5213; Test type: Superiority or Other; p = 0.4822, Mixed Models Analysis; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.30 to 0.64], Standard Error of Mean 0.23

2. Post Hoc Outcome: Brief Pain Index - Item 5, Average Daily Pain Score (Range 0-10) Higher Score Indicates Worse Pain - Per Protocol
Description: Brief pain Index - diabetic painful neuropathy (BPI-DPN) - average daily pain, Item 5 (final 2 day home diary + in clinic assessment at end of 3 week treatment)
Time Frame: 3 weeks of treatment
Population: Per Protocol
Measure: Least Squares Mean (Standard Error); unit: Average daily pain score
Arm/Group | Part 2 - Placebo | Part 2 - Pregabalin + AZD5213 | Part 2 - Pregabalin
Number analyzed (Participants) | 20 | 20 | 20
Average daily pain score | 4.46 (0.45) | 4.35 (0.45) | 4.04 (0.45)
Statistical Analysis 1: Comparison: Part 2 - Pregabalin + AZD5213 vs Part 2 - Pregabalin; Test type: Superiority or Other; p = 0.2237, Mixed Models Analysis; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.20 to 0.82], Standard Error of Mean 0.25 — In direction of Pregabalin
Statistical Analysis 2: Comparison: Part 2 - Placebo vs Part 2 - Pregabalin; Test type: Superiority or Other; p = 0.0978, Mixed Models Analysis; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.93 to 0.08], Standard Error of Mean 0.25 — In direction of Pregabain, positive control
Statistical Analysis 3: Comparison: Part 2 - Placebo vs Part 2 - Pregabalin + AZD5213; Test type: Superiority or Other; p = 0.6610, Mixed Models Analysis; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.62 to 0.40], Standard Error of Mean 0.25

ADVERSE EVENTS:
Time Frame: (5 months)
Description: From start of Part 1 through follow up visit 7 to 14 days after last dose in Part 2, 3 period crossover
Groups:
- Part 1: Part 1 - Pain training + 1 week of single blind placebo
- Overall Study: Overall Study: Part 1 and Part 2
Arm/Group | Part 1 | Part 2 - Placebo | Part 2 - Pregabalin + AZD5213 | Part 2 - Pregabalin | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/30 | 0/28 | 0/30 | 0/83
Other Adverse Events (participants affected / at risk) | 19/83 | 8/30 | 11/28 | 11/30 | 32/83
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (N=83) | Part 2 - Placebo (N=30) | Part 2 - Pregabalin + AZD5213 (N=28) | Part 2 - Pregabalin (N=30) | Overall Study (N=83)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Herper zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic neck pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 5 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Diabetes mellitis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Exotosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopaty (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngael pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days